CLINICAL TRIAL: NCT04440267
Title: A Prospective, Single Arm, Open Label, Clinical Trial to Evaluate the Efficacy of Acute Lymphoblastic Leukemia-Based Therapy in Treating Patients With Acute Leukemia of Ambiguous Lineage
Brief Title: Efficacy of Acute Lymphoblastic Leukemia-Based Therapy in Treating Patients With Acute Leukemia of Ambiguous Lineage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020009
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Acute Leukemia of Ambiguous Lineage
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute | interventions — Vincristine; Daunorubicin; Cyclophosphamide; Asparaginase; Prednisone; Mercaptopurine; Methotrexate; Dexamethasone; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): Patients will receive acute lymphoblastic leukemia (ALL) -based chemotherapy and are permitted to receive allogeneic hematopoietic stem cell transplantation (HSCT) in CR. Otherwise, they will finish the consolidation chemotherapy. Patients with t(9;22) will receive chemotherapy combined with tyrosine kinase inhibitors.
  Interventions: Drug: vincristine; Drug: daunorubicin; Drug: cyclophosphamide; Drug: L-Asparaginase; Drug: prednisone; Drug: mercaptopurine; Drug: methotrexate; Drug: dexamethasone; Drug: Tyrosine kinase inhibitor

INTERVENTIONS:
Drug: vincristine — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: daunorubicin — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: cyclophosphamide — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: L-Asparaginase — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: prednisone — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: mercaptopurine — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: methotrexate — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: dexamethasone — acute lymphoblastic leukemia (ALL) -based chemotherapy
Drug: Tyrosine kinase inhibitor — acute lymphoblastic leukemia (ALL) -based chemotherapy

SUMMARY:
In this prospective, single arm, open label, clinical trial, a total of 50 acute leukemia of ambiguous lineage patients will be enrolled. Patients will receive acute lymphoblastic leukemia (ALL) -based chemotherapy and are permitted to receive allogeneic hematopoietic stem cell transplantation (HSCT) after CR . Otherwise, they will finish the consolidation chemotherapy. Patients with t(9;22) will receive chemotherapy combined with tyrosine kinase inhibitors. The purpose of current study is to evaluate the clinical efficacy of ALL-based chemotherapy，effect of genetic abnormality and minimal residual disease (MRD) on prognosis in patients with acute leukemia of ambiguous lineage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged above 14 years with acute leukemia of ambiguous lineage .
2. Eastern Cooperative Oncology Group (ECOG) Performance status 2.
3. Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal (ULN); serum glutamic-oxaloacetic transaminase(SGOT) and serum glutamic pyruvic transaminase(SGPT) ≤ 2.5 x ULN; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; Patients must have adequate cardiac function (ejection fraction ≥ 45 % on Multiple Gated Acquisition (MUGA) scan).
4. Patients must have the following laboratory values (≥ lower limit of normal (LLN) or corrected to within normal limits with supplements prior to the first dose of study medication.): Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN
5. Patients should sign informed consent form.

Exclusion Criteria:

1. Impaired cardiac function:

   Long QT syndrome or a known family history of long QT syndrome; clinically significant resting brachycardia (<50 beats per minute); ejection fraction < 45 % on MUGA scan. Corrected QT (QTc) interval > 450 msec on baseline ECG (using the QTcF formula). If QTcF interval>450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc. Myocardial infarction within 12 months prior to starting study; other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension, uncontrolled arrhythmias).
2. Other concurrent severe and/or uncontrolled medical conditions:

   Patients with another primary malignant disease, except those that do not currently require treatment; acute or chronic liver, pancreatic or severe renal disease; another severe and/or life-threatening medical disease.
3. Patients who are: (a) pregnant and (b) breast feeding.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 5 years
  From the date of diagnosis until the date of death from any cause,

SECONDARY OUTCOMES:
Relapse free survival (RFS) | up to 5 years
  From the date of CR until the date of relapse or death
The complete remission (CR) rate | up to 2.5 years
  Incidence of complete remission after induction chemotherapy
Mortality within 60 days | up to 60 days
  Proportion of patients died within 60 days

OTHER OUTCOMES:
Chromosomal abnormalities detected by G-banding | Baseline
Fusion genes detected by polymerase chain reaction | Baseline
Mutations detected by next-generation sequencing | Baseline
Minimal residual disease（MRD） | 1 year
  The presence of small numbers of leukemic cells detected by the flow cytometry after remission

CONTACTS AND LOCATIONS:
Locations (1):
- HBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code